CLINICAL TRIAL: NCT05374070
Title: Assessment of Anti-viral Activity of Saliva Obtained From Human Volunteers Following Application of Probiotic Streptococcus Salivarius to the Oral Cavity
Brief Title: Antiviral Activity of Oral Probiotics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: John Hale (Industry)
Responsible Party: Sponsor-Investigator, John Hale, Chief Technology Officer, BLIS Technologies Limited
Organization: BLIS Technologies Limited (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BLTCT2022/2
Record Dates: First submitted 2022-05-09; First posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Lower Respiratory Tract Infection; Upper Respiratory Tract Infection
Keywords: Streptococcus salivarius K12; Probiotic; Antiviral activity; Antibacterial activity; microbial colonization; oral probiotic; powder; prebiotic
MeSH Terms: conditions — Respiratory Tract Infections; Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of the 4 groups consuming powder containing Streptococcus salivarius K12 or S. salivarius M18 with or without prebiotic:
  1. Probiotic Streptococcus salivarius K12 Powder (Dose: 1 Billion cfu/g)
  2. Probiotic Streptococcus salivarius K12 Powder with prebiotic (Dose: 1 Billion cfu/g)
  3. Probiotic Streptococcus salivarius M18 Powder (Dose: 1 Billion cfu/g)
  4. Probiotic Streptococcus salivarius M18 Powder with prebiotic (Dose: 1 Billion cfu/g)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Streptococcus salivarius K12 (Active Comparator): Streptococcus salivarius K12 (Dose 1: 1 Billion colony forming units /g)
  Interventions: Dietary Supplement: Streptococcus salivarius K12 Powder 1 Billion colony forming units /g)
- Streptococcus salivarius K12 with a prebiotic included (Active Comparator): Streptococcus salivarius K12 (Dose 1: 1 Billion colony forming units /g)
  Interventions: Dietary Supplement: Streptococcus salivarius K12 Powder (1 Billion colony forming units /g) with a prebiotic included
- Streptococcus salivarius M18 (Active Comparator): Streptococcus salivarius M18 (Dose 1: 1 Billion colony forming units /g)
  Interventions: Dietary Supplement: Streptococcus salivarius M18 Powder (1 Billion colony forming units /g)
- Streptococcus salivarius M18 with a prebiotic included (Active Comparator): Streptococcus salivarius M18 (Dose 1: 1 Billion colony forming units /g)
  Interventions: Dietary Supplement: Streptococcus salivarius M18 Powder (1 Billion colony forming units /g) with a prebiotic included

INTERVENTIONS:
Dietary Supplement: Streptococcus salivarius K12 Powder 1 Billion colony forming units /g) — Probiotic Streptococcus salivarius K12 products are commercially available in traditional formats such as lozenges for local delivery in the oral cavity to provide oral health benefits. In this study, a powder formulation will be evaluated for its potential of delivering probiotic Streptococcus salivarius K12 to the oral cavity.
  Arms: Streptococcus salivarius K12
Dietary Supplement: Streptococcus salivarius K12 Powder (1 Billion colony forming units /g) with a prebiotic included — In this study, a powder formulation containing Streptococcus salivarius K12 and a prebiotic will be evaluated for its potential of delivering probiotic Streptococcus salivarius K12 to the oral cavity.
  Arms: Streptococcus salivarius K12 with a prebiotic included
Dietary Supplement: Streptococcus salivarius M18 Powder (1 Billion colony forming units /g) — In this study, a powder formulation will be evaluated for its potential of delivering probiotic Streptococcus salivarius M18 to the oral cavity.
  Arms: Streptococcus salivarius M18
Dietary Supplement: Streptococcus salivarius M18 Powder (1 Billion colony forming units /g) with a prebiotic included — In this study, a powder formulation containing S. salivarius M18 and a prebiotic will be evaluated for its potential of delivering probiotic Streptococcus salivarius M18 to the oral cavity.
  Arms: Streptococcus salivarius M18 with a prebiotic included

SUMMARY:
The aim of this study is to test saliva samples obtained from healthy human participants for anti-viral activity after they have consumed S. salivarius probiotic in a powder format.

DETAILED DESCRIPTION:
This is a randomized controlled open pilot study to evaluate saliva samples collected from participants following their consumption of powders containing the commercially marketed probiotic bacterium S. salivarius K12 or S. salivarius M18.

Participants will be randomly assigned to one of the 4 groups consuming probiotic powder containing Streptococcus salivarius K12 or S. salivarius M18 with or without prebiotics (e.g. sugars that may promote probiotic activity). Saliva samples will be collected at predetermined time points pre and post intervention. Antibacterial and Antiviral activity will be determined following established assays. Colonisation efficacy will be determined by enumerating the probiotic in the saliva samples using standard microbiological techniques.

ELIGIBILITY:
Inclusion criteria:

1. In general good health 18 - 80 years of age.
2. Practice good oral hygiene.

Exclusion criteria:

1. Have a history of autoimmune disease or are immunocompromised.
2. Are on concurrent antibiotic therapy or regular antibiotic use within last 1 week
3. History of allergy (e.g. dairy).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-23 (Estimated); Primary Completion 2022-06-23 (Estimated); Study Completion 2022-08-15 (Estimated)

PRIMARY OUTCOMES:
Change in antiviral activity following dosing with probiotic S. salivarius K12 in saliva from Day 0 (baseline) to 3 hours | 3 hours post intervention
  Study will determine the antiviral activity of Streptococcus salivarius K12 without prebiotic in a powder format. The antiviral and antibacterial activity in the saliva will be determined using appropriate assays and Statistical analysis (e.g. Students t-test) will be carried out to compare the participants data for different days (pre and post time points) and different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g Microsoft Excel).
Change in antiviral activity following dosing with probiotic S. salivarius K12 in saliva from Day 0 (baseline) to 8 hours | 8 hours post intervention
  Study will determine the antiviral activity of Streptococcus salivarius K12 without prebiotic in a powder format. The antiviral and antibacterial activity in the saliva will be determined using appropriate assays and Statistical analysis (e.g. Students t-test) will be carried out to compare the participants data for different days (pre and post time points) and different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g Microsoft Excel).
Change in antiviral activity following dosing with probiotic S. salivarius K12 with prebiotic in saliva from Day 0 (baseline) to 3 hours | 3 hours post intervention
  Study will determine the antiviral activity of Streptococcus salivarius K12 with prebiotic in a powder format. The antiviral and antibacterial activity in the saliva will be determined using appropriate assays and Statistical analysis (e.g. Students t-test) will be carried out to compare the participants data for different days (pre and post time points) and different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g Microsoft Excel).
Change in antiviral activity following dosing with probiotic S. salivarius K12 with prebiotic in saliva from Day 0 (baseline) to 8 hours | 8 hours post intervention
  Study will determine the antiviral activity of Streptococcus salivarius K12 with prebiotic in a powder format. The antiviral and antibacterial activity in the saliva will be determined using appropriate assays and Statistical analysis (e.g. Students t-test) will be carried out to compare the participants data for different days (pre and post time points) and different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g Microsoft Excel)
Change in antiviral activity following dosing with probiotic S. salivarius M18 in saliva from Day 0 (baseline) to 3 hours | 3 hours post intervention
  Study will determine the antibacterial activity of Streptococcus salivarius M18 without prebiotic in a powder format. The antibacterial activity in the saliva will be determined using appropriate assays and Statistical analysis (e.g. Students t-test) will be carried out to compare the participants data for different days (pre and post time points) and different formulations with the level of significance of p≤0.05.
Change in antiviral activity following dosing with probiotic S. salivarius M18 in saliva from Day 0 (baseline) to 8 hours | 8 hours post intervention
  Study will determine the antibacterial activity of Streptococcus salivarius M18 without prebiotic in a powder format. The antibacterial activity in the saliva will be determined using appropriate assays and Statistical analysis (e.g. Students t-test) will be carried out to compare the participants data for different days (pre and post time points) and different formulations with the level of significance of p≤0.05.
Change in antiviral activity following dosing with probiotic S. salivarius M18 with prebiotic in saliva from Day 0 (baseline) to 3 hours | 3 hours post intervention
  Study will determine the antibacterial activity of Streptococcus salivarius M18 with prebiotic in a powder format. The antibacterial activity in the saliva will be determined using appropriate assays and Statistical analysis (e.g. Students t-test) will be carried out to compare the participants data for different days (pre and post time points) and different formulations with the level of significance of p≤0.05.
Change in antiviral activity following dosing with probiotic S. salivarius M18 with prebiotic in saliva from Day 0 (baseline) to 8 hours | 8 hours post intervention
  Study will determine the antibacterial activity of Streptococcus salivarius M18 with prebiotic in a powder format. The antibacterial activity in the saliva will be determined using appropriate assays and Statistical analysis (e.g. Students t-test) will be carried out to compare the participants data for different days (pre and post time points) and different formulations with the level of significance of p≤0.05.

CONTACTS AND LOCATIONS:
Overall Officials: John D Hale, PhD, Study Director — Blis Technologies Ltd, Dunedin, New Zealand; John R Tagg, PhD, Principal Investigator — Blis Technologies Ltd, Dunedin, New Zealand; Liam Harold, PhD, Principal Investigator — Blis Technologies Ltd, Dunedin, New Zealand
Locations (1):
- Blis Technologies Ltd, Dunedin, Otago, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Data information and information included in the protocol and the Clinical study report will be shared to other researchers and/or in publications in due course.
Supporting Information: Study Protocol, CSR
Time Frame: Study report 3 months after the completion of the study.
Access Criteria: Summary study report will be shared by Principal investigator upon request if not published in public literature.

REFERENCES:
- [Background] Hyink O, Wescombe PA, Upton M, Ragland N, Burton JP, Tagg JR. Salivaricin A2 and the novel lantibiotic salivaricin B are encoded at adjacent loci on a 190-kilobase transmissible megaplasmid in the oral probiotic strain Streptococcus salivarius K12. Appl Environ Microbiol. 2007 Feb;73(4):1107-13. doi: 10.1128/AEM.02265-06. Epub 2006 Dec 28. PMID 17194838
- [Background] Burton JP, Chilcott CN, Wescombe PA, Tagg JR. Extended Safety Data for the Oral Cavity Probiotic Streptococcus salivarius K12. Probiotics Antimicrob Proteins. 2010 Oct;2(3):135-44. doi: 10.1007/s12602-010-9045-4. PMID 26781236